CLINICAL TRIAL: NCT02516787
Title: Coherence Between Brain Cortical Function and Neurocognitive Performance During Changed Gravity Conditions
Acronym: CORTICOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10-082
Record Dates: First submitted 2015-07-28; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EEG and NIRS measurements (Other)
  Interventions: Other: Parabolic flight; Other: EEG measurement; Other: NIRS measurements

INTERVENTIONS:
Other: Parabolic flight
Other: EEG measurement — Electro cortical power in alpha frequency ranges (EEG-LORETA)
Other: NIRS measurements — Brain tissue oxygenation ( oxy- or deoxygenated hemoglobin values) - NIRS

SUMMARY:
Alongside a well-known physiological deconditioning, such as a decrease in muscle mass or bone demineralization, extended stays in weightlessness also cause cognitive dysfunction. However, the studies on this subject during space missions short or long term could not determine how these cognitive dysfunction resulted from a direct effect of weightlessness or a stress-related effect.

Analysis of electro-encephalography (EEG) using a standardized mapping method is used to study the changes of operation of the cerebral cortex as the near infrared spectroscopy (NIRS) is a reflection of changes in the cerebral hemodynamics. Their combined use is a relatively simple and economical method for studying brain changes in an environment where the normal brain imaging techniques can not be used.

The main objective of this experiment is to evaluate the alterations in brain cortical activity and brain oxygenation level induced by micro- and hypergravity conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (men or women),
* aged from 18 to 65,
* affiliated to a Social Security system and, for non-French resident, holding an European Health Insurance Card (EHIC)
* who accept to take part in the study,
* who have given their written stated consent,
* who already participated in parabolic flights (even in the same campaign)
* All subjects will pass a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Exclusion Criteria:

* Persons who took part in a previous biomedical research protocol, of which exclusion period is not terminated,
* Persons with prior serious injuries to their head
* Persons who take any medication or drugs influencing their central nervous system or cognitive performance
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
alterations in brain cortical activity (EEG) | baseline
brain oxygenation level (NIRS) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France